CLINICAL TRIAL: NCT07343141
Title: A Prospective, Randomized, Evaluator/Subject-blinded, Single-center, Split-Face Controlled Clinical Study: To Evaluate the Safety and Efficacy of Poly-L-lactic Acid Implants for the Correction of Nasolabial Folds
Brief Title: To Evaluate the Safety and Efficacy of Poly-L-lactic Acid Implants for the Correction of Nasolabial Folds
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SciVision Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RDCT-NFFU
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Nasolabial Fold Correction
Keywords: Poly-L-lactic Acid; Nasolabial folds

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FUYANMEI Poly-L-Lactic Acid (Experimental): Poly-L-Lactic Acid
  Interventions: Device: FUYANMEI Poly-L-Lactic Acid
- Sculptra® (Active Comparator): Poly-L-Lactic Acid
  Interventions: Device: Sculptra®

INTERVENTIONS:
Device: FUYANMEI Poly-L-Lactic Acid — Poly-L-Lactic Acid
  Arms: FUYANMEI Poly-L-Lactic Acid
Device: Sculptra® — Poly-L-Lactic Acid
  Arms: Sculptra®

SUMMARY:
The goal of this clinical trial is to evaluate the safety and effectiveness of a poly-L-lactic acid (PLLA) dermal implant for the correction of nasolabial folds. The study also aims to determine whether the investigational product (FUYANMEI Poly-L-Lactic Acid) is non-inferior to the control product (Sculptra).

The main questions it aims to answer are:

* Is the effectiveness rate based on the Wrinkle Severity Rating Scale (WSRS) at 6 months after injection for the investigational group non-inferior to that of the control group?
* How does the investigational product perform in terms of global aesthetic improvement as assessed by blinded evaluators and by subjects?
* What is the safety profile of the investigational product, including the incidence, severity, and relatedness of adverse events (AEs), serious adverse events (SAEs), and device deficiencies (DDs)?

Researchers will compare the investigational PLLA implant to an approved PLLA implant using a prospective, randomized, evaluator- and subject-blinded, single-center, split-face controlled study design. Approximately 121 eligible participants will be enrolled.

Participants will:

* Receive treatment with the investigational product and the control product according to the split-face design
* Be followed for 24 months after injection
* Return to the clinic at 1, 3, 6, 12, 18, and 24 months post-injection for follow-up visits
* Undergo blinded evaluator assessments of WSRS and Global Aesthetic Improvement Scale (GAIS)
* Complete subject self-assessments of GAIS and treatment satisfaction
* Be monitored throughout the study for adverse events, serious adverse events, and medical device deficiencies

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent prior to any study-specific procedures.
2. Male or female subjects aged between 19 and 65 years.
3. Presence of bilateral nasolabial fold wrinkles with a Wrinkle Severity Rating Scale (WSRS) score of moderate (Grade 3) or severe (Grade 4) at baseline.
4. Willingness and ability to comply with all protocol-required follow-up visits and procedures.

Exclusion Criteria:

1. History of hypertrophic scarring or keloid formation.
2. Presence of active infection or dermatologic conditions at or near the intended injection site that may interfere with the evaluation.
3. Underwent major surgery within 3 months prior to study initiation.
4. Diagnosed with autoimmune diseases, malignancies, psychiatric disorders, or poorly controlled chronic medical conditions.
5. Prior treatment with or planned use of permanent dermal fillers at the intended injection site.
6. Prior treatment with or planned use of temporary fillers, collagen stimulators, or thread lifting at the injection site within 12 months prior to screening or during the study period.
7. Underwent or plans to undergo laser treatments to the mid- or lower face within 3 months prior to treatment or during the study period.
8. Underwent or plans to undergo ultrasound or radiofrequency skin tightening procedures to the mid- or lower face within 6 months prior to treatment or during the study period.
9. Known hypersensitivity to poly-L-lactic acid or any components of the investigational device, or any other significant allergy as deemed by the investigator to pose risk to the subject.
10. Planned surgeries or medications during the study period that may cause significant weight changes.
11. Pregnant or breastfeeding women, or women intending to become pregnant during the study period.
12. Participation in another interventional clinical trial that has not concluded within 30 days prior to screening, or plans to participate in another interventional clinical study during the course of this study.
13. Any other condition or situation that, in the opinion of the investigator, renders the subject unsuitable for study participation.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
The responder rate based on the Wrinkle Severity Rating Scale (WSRS). | at Month 6 post-injection
  The WSRS responder rate at Month 6 post-injection was compared between the treatment and control groups. A WSRS responder was defined as a participant who achieved an improvement of at least 1 point in the WSRS score compared with baseline.

SECONDARY OUTCOMES:
Wrinkle Severity Rating Scale (WSRS) scores | at baseline, immediately post-treatment (Day 0), and at Months 1, 3, 6, 12, 18, and 24 post-injection
  WSRS was assessed using a 5-point scale (1-5), with higher scores indicating greater wrinkle severity. Blinded evaluators assessed WSRS scores at baseline, immediately post-treatment (Day 0), and at Months 1, 3, 6, 12, 18, and 24 following injection.
WSRS responder rates | at baseline, Day 0, and Months 1, 3, 12, 18, and 24 post-injection
  WSRS responder rates assessed by blinded evaluators at baseline, Day 0, and Months 1, 3, 12, 18, and 24 post-injection. A WSRS responder was defined as a participant who achieved an improvement of at least 1 point in the WSRS score compared with baseline.
Change in nasolabial fold volume | at baseline, Day 0, and Months 1, 3, 6, 12, 18, and 24 post-injection
  Images were captured using a VECTRA H2 3D camera (Canfield Scientific) at a fixed distance from the subject's face under standardized lighting and background conditions. The resulting image files were analyzed for volumetric measurements using 3D imaging software. Changes in nasolabial fold volume from baseline (Day 0) were assessed at Months 1, 3, 6, 12, 18, and 24 using the three-dimensional imaging system.
Global Aesthetic Improvement Scale (GAIS) scores | at immediately post-treatment (Day 0), and Months 1, 3, 6, 12, 18, and 24 post-injection
  GAIS scores were measured using a 5-point scale (1-5), with lower scores indicating poorer improvement. Blinded evaluators assessed GAIS scores immediately post-treatment (Day 0) and at Months 1, 3, 6, 12, 18, and 24 after injection.
Subject-reported GAIS scores | at immediately post-treatment (Day 0), and Months 1, 3, 6, 12, 18, and 24 post-injection
  Subject-reported GAIS scores at immediately post-treatment (Day 0), and Months 1, 3, 6, 12, 18, and 24 post-injection.
Subject-reported satisfaction scores | at Months 1, 3, 6, 12, 18, and 24 post-injection
  Subject-reported satisfaction was assessed at Months 1, 3, 6, 12, 18, and 24 post-injection. Participants rated their satisfaction with the treatment's safety and effectiveness using a questionnaire scored on a 5-point scale (1-5), where 5 indicated very high satisfaction and 1 indicated very low satisfaction.
Incidence of Adverse Events (AEs) | at Day 0, Months 1, 3, 6, 12, 18, and 24 post-injection
  The incidence rate of adverse events (AEs), expressed as a percentage, will be calculated based on subjects who reported AEs or whose AEs were observed by investigators. The incidence rate will be determined using the following formula: AE (%) = (number of subjects who experienced AEs in each group ÷ total number of subjects in each group) × 100. Adverse events will be assessed on the day of treatment and at Months 1, 3, 6, 12, 18, and 24 post-treatment.
Incidence of Serious Adverse Events (SAEs) | at Day 0, Months 1, 3, 6, 12, 18, and 24 post-injection
  The incidence rate of serious adverse events (SAEs), expressed as a percentage, will be calculated based on subjects who reported SAEs or whose SAEs were observed by investigators. The incidence rate will be determined using the following formula: SAE (%) = (number of subjects who experienced SAEs in each group ÷ total number of subjects in each group) × 100. Adverse events will be assessed on the day of treatment and at Months 1, 3, 6, 12, 18, and 24 post-treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided